CLINICAL TRIAL: NCT06225271
Title: Effects of the Combined Intervention of Exercise, Fruit, and Vitamin Supplementation on Frailty in Older Adults: A Cohort-based Cluster- Randomized Controlled Trial
Brief Title: Effects of the Combined Intervention of Exercise, Fruit, and Vitamin Supplementation on Frailty in Older Adults
Acronym: EFVF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Collaborators: Suzhou Center for Disease Control and Prevention (Unknown)
Responsible Party: Principal Investigator, Chong Shen, Professor, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GSKY20230103
Record Dates: First submitted 2023-12-22; First posted 2024-01-25 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-09

CONDITIONS: Frailty
Keywords: Older adults; Frailty; Exercise; Fruit; Vitamin supplementation; Cluster- randomized controlled trial; Muscle loss
MeSH Terms: conditions — Frailty; Motor Activity; Muscular Atrophy | interventions — Fruit

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group will receive group intervention and individual intervention. Group interventions will include participants' communication meeting and other approach, such as self-management group. They will also receive the combined intervention of physical activity, fruit, and vitamin supplementation 3 times a week for 2 months (the 1st and 6th months).
  Interventions: Behavioral: the combined intervention of exercise, fruit, and vitamin supplementation
- Control group (No Intervention): Participants in the control arm will not receive any intervention.

INTERVENTIONS:
Behavioral: the combined intervention of exercise, fruit, and vitamin supplementation — Group intervention
  After each intervention, investigators will hold a 15-minute communication and discussion session for the participants. Besides, community health workers will organize at least one health education activity per week during the intervention for no less than 45 minutes.
  Individual intervention
  Physical activity
  The participants will be gathered at the community activity center or day care center. The participants will be allowed to exercise in a way that interests them. The duration of exercise should be longer than 30 minutes.
  Fruit supplementation
  Consideration of seasonal supply situation and the participants' diabetic status, various types of fruit will be prepared. The fruit will be divided into 50g/100g servings. Participants will be required to eat on site.
  Vitamin supplementation
  During the intervention, the participants will be required to take 1 tablet of vitamin B complex plus 1 tablet of vitamin C every day.
  Arms: Intervention group

SUMMARY:
The goal of this cohort-based cluster-randomized controlled trial is to investigate the effect of the combined intervention of exercise, fruit, and vitamin supplementation on frailty among older adults. Older individuals aged 65~80 years old with low physical activity levels and low fruit intake will be recruited. 14 clusters will be randomized into 2 arms with 1:1 ratio. Participants in the intervention arm will receive the combined intervention of physical activity, fruit, and vitamin supplementation 3 times a week for 2 months (the 1st and 6th months). They will also be given group interventions, such as self-management group activity or health education, at least once a week. Participants in the control arm will not receive any intervention.

DETAILED DESCRIPTION:
Objectives Primary objectives

• To evaluate the effect of the combined intervention of exercise, fruit, and vitamin supplementation on preventing muscle loss among older adults over the 12-month period.

Secondary objectives

* To evaluate the effect of the combined intervention of exercise, fruit, and vitamin supplementation on preventing muscle loss in older adults over 6 months.
* To evaluate the effect of the combined intervention of exercise, fruit, and vitamin supplementation on ameliorating frailty in older adults over 6 and 12 months.
* To evaluate the effect of the combined intervention of exercise, fruit, and vitamin supplementation on improving healthy behavior of physical activity and fruit intake in older adults over 12 months.
* To evaluate the effect of the combined intervention of exercise, fruit, and vitamin supplementation on lower the risk of all-cause hospitalization in the older adults over 12 months.
* To evaluate the effect of the combined intervention of exercise, fruit, and vitamin supplementation on lower the risk of all-cause death, cardiovascular and cerebrovascular disease in the older adults over 12 and 24 months.
* To evaluate the effect of the combined intervention of exercise, fruit, and vitamin supplementation on regulating blood lipids in the older adults over 12 and 24 months.
* To evaluate the effect of the combined intervention of exercise, fruit, and vitamin supplementation on regulating blood glucose in the older adults over 12 and 24 months.
* To evaluate the health economic effectiveness of the combined intervention of exercise, fruit, and vitamin supplementation.

Sample size

Sample size was estimated using the Power Analysis and Sample Size (PASS) software (version 15.0.5) based on data from published research. Previous studies showed that the Cohens' d value was between 0.18~1.78. With these data, we estimated effect size of Cohen' d = 0.45, considering probabilities of 5% for type I error, 20% for type II error, and 0.05 for intraclass correlation coefficient (ICC). We randomized all 14 clusters (villages) into two arms with 1:1 ratio, and the total sample size was calculated to be 700 (50 participates per cluster). A conservative estimate of 25% loss to follow-up or drop-out indicates a total of 934 participates is needed.

ELIGIBILITY:
Inclusion Criteria:

1. Permanent resident population aged 65~80 years;
2. Able to walk independently indoors and outdoors;
3. Physical activity less than 1400 metabolic equivalent task (MET)-min/week and fruit intake less than 50 g/day；
4. Have not taken vitamin B and vitamin C supplementation in the past 3 months.

Exclusion Criteria:

1. Presence of a history of fracture;
2. Patients with severe impairment of renal or hepatic fuction. Severe hepatic impairment is defined as serum alanine aminotransferase and aspartate aminotransferase levels above 100 U/L, while severe renal impairment is defined as estimated glomerular filtration rate (eGFR) < 45 mL/min, calculated according to the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equations.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 934 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
The change in handgrip strength at 12 months from baseline. | Baseline and 12 months
  Handgrip strength will be measured using a hand-held grip dynamometer. Participants will be asked to grip the dynamometer with left hand and right hand respectively while standing, maintaining their arm close to the body and straight down, exerting maximum force. This test will be conducted 3 times, and the values will be recorded in kilograms.

SECONDARY OUTCOMES:
The change in handgrip strength at 6 months from baseline. | Baseline and 6 months
  Handgrip strength will be measured using a hand-held grip dynamometer. Participants will be asked to grip the dynamometer with left hand and right hand respectively while standing, maintaining their arm close to the body and straight down, exerting maximum force. This test will be conducted 3 times, and the values will be recorded in kilograms.
The change in frailty index at 6 months and 12 months from baseline. | Baseline, 6 months, and 12 months
  Outcome is defined as the change in the score of modifiable variables in the frailty index from baseline. The frailty index consisted 28 variables covering age, physical measurement, sleep quality, history of surgery, fall, and fracture, history of the disease, oral hygiene, respiratory function, and physical function self-assessment aspects. 24 of the 28 variables can be changed. The frailty index is a continuous variable that ranged from 0 to 33, with a higher value indicating a worse, frailer status.
The change in the quantity and frequency of fruit intake at 12 months from baseline. | Baseline and 12 months
  Fruit intake will be collected by questionnaire for the frequency of consumption and weights per intake. The frequency will be determined by filling in the number of times the participants eat fruit per week/day/monthly/year. Fruit quantity is determined by the product of frequency and weights of a single fruit intake.
The change in physical activity volume and intensity at 12 months from baseline. | Baseline and 12 months
  Information on physical activity levels during the past week will be collected through the International Physical Activity Questionnaire Scale-Short Form (IPAQ-SF). The IPAQ-SF captures four levels of physical activity intensity: vigorous-intensity physical activity, moderate-intensity physical activity, walking time, and average sitting time on weekdays, including sedentary work. Physical activity volume will be determined by summing the metabolic equivalent task (MET)-min/week values for walking, moderate physical activity, and vigorous physical activity. Higher values represent higher levels of physical activity, with a minimum value of 0.
The incidence of a composite of all-cause death, cardiovascular and cerebrovascular diseases over 12 and 24 months. | 12 months, and 24 months
The incidence of all-cause death over 12 and 24 months. | 12 months, and 24 months
The incidence of cardiovascular and cerebrovascular diseases over 12 and 24 months. | 12 months, and 24 months
The change in low-density lipoprotein cholesterol (LDL-C) at 12 months and 24 months from baseline. | Baseline, 12 months, and 24 months
The change in high density lipoprotein cholesterol (HDL-C) at 12 months and 24 months from baseline. | Baseline, 12 months, and 24 months
The change in total cholesterol (TC) at 12 months and 24 months from baseline. | Baseline, 12 months, and 24 months
The change in triglycerides (TG) at 12 months and 24 months from baseline. | Baseline, 12 months, and 24 months
The change in fasting blood glucose at 12 months and 24 months from baseline. | Baseline, 12 months, and 24 months
Incremental cost-effectiveness ratio (ICER) | Baseline and 12 months
  The outcome defined as the excess cost of a strategy over the cost of the baseline strategy divided by the incremental difference in effectiveness between the strategy in question and the baseline strategy.

CONTACTS AND LOCATIONS:
Locations (1):
- Suzhou Center for Disease Control and Prevention, Suzhou, Jiangsu, China

REFERENCES:
- [Result] Scheinin TM. [Rupture of the left main bronchus and pulmonary artery caused by subcutaneous thoracic injuries]. Thoraxchir Vask Chir (1962). 1966 Feb;14(1):54-6. doi: 10.1055/s-0028-1100774. No abstract available. German. PMID 5234793
- [Result] Gomes GS. [Sauna]. Rev Bras Med. 1970 Jan;27(1):47-9. No abstract available. Portuguese. PMID 5517808
- [Result] Inaba Y, Tanaka Y, Ishii S, Morimoto T, Sato K. Ibaraki virus, an agent of epizootic disease of cattle resembling bluetongue. IV. Physicochemical and serological properties of the virus. Jpn J Microbiol. 1970 Sep;14(5):351-60. doi: 10.1111/j.1348-0421.1970.tb00535.x. No abstract available. PMID 4319727
- [Result] Kwon J, Yoshida Y, Yoshida H, Kim H, Suzuki T, Lee Y. Effects of a combined physical training and nutrition intervention on physical performance and health-related quality of life in prefrail older women living in the community: a randomized controlled trial. J Am Med Dir Assoc. 2015 Mar;16(3):263.e1-8. doi: 10.1016/j.jamda.2014.12.005. Epub 2015 Feb 3. PMID 25659620
- [Result] Chen B, Li M, Zhao H, Liao R, Lu J, Tu J, Zou Y, Teng X, Huang Y, Liu J, Huang P, Wu J. Effect of Multicomponent Intervention on Functional Decline in Chinese Older Adults: A Multicenter Randomized Clinical Trial. J Nutr Health Aging. 2023;27(11):1063-1075. doi: 10.1007/s12603-023-2031-9. PMID 37997729

DOCUMENTS (2):
  • Study Protocol (2024-01-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT06225271/Prot_000.pdf
  • Statistical Analysis Plan (2025-09-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT06225271/SAP_001.pdf